CLINICAL TRIAL: NCT00953810
Title: RandomiZed AmbulatOry Interventional ProgrAm in Heart Failure PatieNts (ZOPAN)
Brief Title: Educational Intervention in Heart Failure Patients
Acronym: ZOPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Tomasz M. Rywik MD,Ph.D., Institute of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7/115/2003/101/1304
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Heart Failure
Keywords: heart failure; education; non-pharmacological management; prognosis
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): General heart failure population staying under regular care of their primary care physician
- Intervention (Active Comparator): Like control plus one education training regarding heart failure aspects and management
  Interventions: Other: Educational training regarding heart failure

INTERVENTIONS:
Other: Educational training regarding heart failure — Like control plus one education training regarding heart failure aspects and management
  Other Names: education
  Arms: Intervention

SUMMARY:
The main aim of this randomized study was to evaluate the effect of educational intervention on patients with heart failure and their care-giver with regard to patients' prognosis.

DETAILED DESCRIPTION:
Part I: This is a multicenter study on the effect of educational intervention on heart failure patients and their caregivers with respect to patients' prognosis, social support and quality of life. Subsequent patients with heart failure (based on the inclusion criteria) coming to selected, ambulatory physician, were randomized to either a control or intervention group. Both groups underwent questionnaire evaluation regarding clinical assessment and evaluation of familiarity with aspects of heart failure along with social support and quality of life. Clinical assessment included information on demography, social status, medical history, pharmacotherapy, diagnostic procedures, and utilization of health system resources. After recruitment, patients from intervention group and their caregivers underwent one educational training, during which they received materials on the management of heart failure. Before the meeting, data on familiarity with heart failure were acquired from patients' relatives. During further follow up all participants stayed under regular care from their ambulatory physicians. After 6 months patients underwent short term evaluation based on designated questionnaires, with special attention paid to hospitalization and ambulatory visits due to heart failure. Also data on heart failure knowledge, social support and quality of life was collected. Without any further intervention, follow up was continued. Next long term assessment was undertaken after approximately 3 years from the recruitment. As previously patients fulfilled questionnaires regarding information on their familiarity with heart failure management and social support as well as quality of life. Primary end points of the study were: death, hospitalization (including cardiovascular hospitalizations) and ambulatory visits. Secondary end points included social support and quality of life.

Sub-study: genetic polymorphism - blood specimens collected during one of the visits and stored for further evaluation in future. Study population - all main study participants who gave their informed consent to this part of protocol. Aims: to describe the potential of selected genes candidates polymorphism on the heart failure prognosis and survival in patients NYHA class II-IV.

ELIGIBILITY:
Inclusion Criteria

* Symptoms of heart failure
* EF < 45% (during past 2 years) or abnormal ECG and chest x-ray when echo unavailable
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Severe COPD
* Serious comorbidities, influencing life expectancy or quality of life
* Alcohol and drug addict
* Post MI less than 6 months
* Dementia
* Living in home nursing facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2004-04; Primary Completion 2007-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Primary end points of the study were: death, hospitalization (including cardiovascular hospitalisation)and ambulatory visits. | 6 months and 3 years

SECONDARY OUTCOMES:
Secondary end points included social support and quality of life. | 6 months and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M Rywik, MD, Study Director — Heart Failure and Transplantology Department Institute of Cardiology; Jerzy Korewicki, Md, Ph.D, Principal Investigator — Heart Failure and Transplantology Department; Wojciech Drygas, MD, Ph.D, Principal Investigator — Department of Cardiovascular Epidemiology and Prevention Institute of Cardiology; Grażyna Broda, MD, Ph.D, Principal Investigator — Department of Cardiovascular Epidemiology and Prevention Institute of Cardiology
Locations (10):
- Poland (10):
  - Heart Failure and Transplantology Department Institute of Cardiology, Warsaw, Alpejska 42
  - Oddział Kardiologiczny Szpital Wojewódzki, Ciechanów
  - - Klinika Chorób Wewnętrznych I Rehabilitacji Kardiologicznej, Gdansk
  - Oddział Wewnętrzny Szpital Rejonowy, Grójec
  - Oddział Kardiologii Szpital Wojewódzki, Koszalin
  - - KATEDRA CHORÓB WEWNĘTRZNYCH i GERONTOLOGII, Krakow
  - Oddział Kardiologiczno-Internistyczny Miejski Szpital Zespolony, Olsztyn
  - Ii Klinika Kardiologii A.M, Poznan
  - Oddział Kardiologiczny Radomski Szpital Specjalistyczny, Radom
  - Oddział Kardiologiczny Samodzielny Specjalistyczny Szpital Wojewódzki, Siedlce

REFERENCES:
- [Derived] Rywik TM, Kolodziej P, Targonski R, Fedyk-Lukasik M, Nowicka A, Zinka E, Zbyszynski B, Achremczyk P, Gorski J, Muder A, Sadowski J, Leszek P, Kurjata P, Broda G, Korewicki J. Characteristics of the heart failure population in Poland: ZOPAN, a multicentre national programme. Kardiol Pol. 2011;69(1):24-31. PMID 21267960